CLINICAL TRIAL: NCT06050590
Title: Impact of Peripheral Sensory Stimulation of the Hand and Synchronized Deep Breathing in the Treatment of Post-Traumatic Stress Disorder: Assessing Safety and Effectiveness
Brief Title: NeuroGlove PTSD Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NeuroGlove LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REG-1003
Record Dates: First submitted 2023-07-17; First posted 2023-09-22 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2023-09

CONDITIONS: PTSD; Post Traumatic Stress Disorder
Keywords: PTSD; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: NeuroGlove
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- NeuroGlove Treatment Arm (Experimental): Study participants undergoing treatment using the NeuroGlove.
  Interventions: Device: NeuroGlove

INTERVENTIONS:
Device: NeuroGlove — Study participant with PTSD will undergo daily at home treatment using the NeuroGlove.

SUMMARY:
This is a prospective, home-based, interventional clinical study in which 6 subjects will be enrolled. Six (6) subjects who suffer from post-traumatic stress disorder will receive treatment using the NeuroGlove.

DETAILED DESCRIPTION:
This is a prospective, home-based, interventional clinical study in which 6 subjects will be enrolled. Six (6) subjects who suffer from post-traumatic stress disorder will receive treatment using the NeuroGlove.

There will be a single cohort in the study consisting of the subjects with PTSD who will receive treatment with NeuroGlove.

The trial is intended to evaluate the impact of the device use on active PTSD symptoms and subject sense of well-being.

ELIGIBILITY:
Inclusion Criteria:

* Able to and willing to provide informed consent. Legally authorized representatives (LARs) will not be allowed to consent on behalf of the subject.
* Men and women ≥18 and <85 years of age.
* Carry an active diagnosis of PTSD.
* Suffer from PTSD symptoms that impact subject's daily activities and quality of life.

Exclusion Criteria:

* Physical limitations of the upper extremity (e.g., fracture, joint deformity, severe spasticity/contracture, wounds, skin breakdown, lymphedema, etc.)
* Subject lacks the ability to comprehend or following instructions, or for any reason, in the opinion of the investigator, would be unlikely or unable to comply with study protocol requirements.
* Currently participating in another interventional clinical trial. (Observational clinical trial participation is allowed for study enrollment.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-08-27 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
PTSD Symptom Reduction | 4 weeks
  Change in PTSD symptoms and subject's sense of well-being
Portion of participants with adverse events | 4 weeks
  Rate and severity of adverse events related to the use of the NeuroGlove.

SECONDARY OUTCOMES:
PTSD Symptom Severity | 4 weeks
  Change in severity of symptoms related to PTSD using NSESSS

CONTACTS AND LOCATIONS:
Overall Officials: Eric Nussbaum, MD, Principal Investigator — NeuroGlove LLC
Locations (1):
- NeuroGlove, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
The data will only be used by the sponsor organization and investigators.